CLINICAL TRIAL: NCT06860815
Title: Pilot Study of Cemiplimab and Hepatic Radioembolization in Patients With Liver Dominant Metastatic Breast Cancer
Brief Title: Cemiplimab and Transarterial Radioembolization With Y-90 SIR-S Spheres for the Treatment of Liver Directed Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23768; NCI-2025-00340 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23768 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-02-04; First posted 2025-03-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Carcinoma in the Liver
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy; Specimen Handling; cemiplimab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cemiplimab, Y90 SIR-Spheres, TARE) (Experimental): Patients receive cemiplimab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive Y90 SIR-Spheres intratumorally via TARE over 60-90 minutes once during days 7-14 and on day 67. Patients also undergo tumor biopsy at baseline and at day 42 after immunotherapy begins. Additionally patients also undergo blood sample collection and CT or MRI throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Biological: Cemiplimab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Radiation: Transarterial Radioembolization; Radiation: Yttrium Y 90 Resin Microspheres

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Cemiplimab — Given IV
  Other Names: Cemiplimab RWLC; Cemiplimab-rwlc; Libtayo; REGN 2810; REGN-2810; REGN2810
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Transarterial Radioembolization — Undergo TARE
  Other Names: Hepatic Radioembolization; TARE; Transarterial Hepatic Radioembolization
Radiation: Yttrium Y 90 Resin Microspheres — Given intratumorally
  Other Names: SIR-Spheres; Y-90 Sirsphere

SUMMARY:
This phase II trial tests how well cemiplimab and transarterial radioembolization (TARE) with yttrium-90 (Y90) SIR-Spheres, registered trademark, works in treating breast cancer that has spread from where it first started (primary site) to the liver (metastatic). Immunotherapy with monoclonal antibodies, such as cemiplimab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. TARE is a treatment that uses radioactive microspheres, such as Y90 SIR-S Spheres, to both cause hepatic artery embolization and to deliver regional radiotherapy. Y90 SIR-S Spheres is an injectable form of the radioisotope yttrium Y 90 encapsulated in resin microspheres. When injected into the artery supplying the tumor, yttrium Y 90 resin microspheres block the tumor blood vessels and deliver the yttrium Y 90 directly to the tumor site, which may kill or slow tumor growth. Giving cemiplimab and Y90 SIR-Spheres by TARE to the tumor in the liver may kill more tumor cells in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the effect of cemiplimab and yttrium Y90 resin microspheres (90Y TARE) on immune activation in the treated tumor based on CD8+ T cells.

SECONDARY OBJECTIVES:

I. To evaluate other measures of changes (both in treated and untreated lesions after the first TARE treatment) in the tumor microenvironment (TME) of 10 metastatic breast cancer (MBC) patients with liver-dominant disease.

II. To identify systemic immune activation in the peripheral blood. III. To determine the safety and tolerability of cemiplimab and hepatic radioembolization in patients with liver dominant metastatic breast cancer using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 criteria.

IV. To evaluate objective tumor response of the target lesion treated with Y90 by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST (mRECIST).

OUTLINE:

Patients receive cemiplimab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients receive Y90 SIR-Spheres intratumorally via TARE over 60-90 minutes once during days 7-14 and on day 67. Patients also undergo tumor biopsy at baseline and at day 42 after immunotherapy begins. Additionally patients also undergo blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 3 months within 1 year of start of treatment, and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Must have a life expectancy of at least 12 weeks
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy)
* Male patients must be surgically sterile, or if sexually active and having a pre-menopausal female partner then must be using an acceptable form of contraception
* Patients with metastatic breast cancer, previously treated with ≥ 1 line of chemotherapy in metastatic setting
* Candidate for TARE based on evaluation by board certified interventional radiologist; must have measurable metastatic liver disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as outlined in RECIST version 1.1; not all liver tumors will be treated with TARE in a single session
* Liver tumor burden < 50%
* No radiographic or clinical evidence of cirrhosis
* Other treated stable metastases are allowed, including treated stable brain metastases
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Body weight > 30 kg
* No untreated, active hepatitis
* Hemoglobin ≥ 9.0 g/dL (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Absolute neutrophil count (ANC) ≥ 1500/uL (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Platelet count ≥ 75000/uL (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Total bilirubin < 2.0mg/dL (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT/serum glutamic pyruvic transaminase [SGPT]) ≤ 5 x upper limit of normal (ULN) (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Albumin ≥ 2.8 g/dL (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* International normalized ration (INR) ≤ 1.6 (within 14 days prior to day 1 of protocol therapy unless otherwise stated)
* Measured creatinine clearance (CL) > 40 mL/min or calculated creatinine CL > 40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance (within 14 days prior to day 1 of protocol therapy unless otherwise stated)

Exclusion Criteria:

* Prior immunotherapy in the past 12 months
* Progressing or untreated extra-hepatic metastatic disease
* Autoimmune disease requiring therapy; immunodeficiency, or any disease process requiring immunosuppressive therapy
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Portal vein invasion
* Evidence of diffuse metastatic disease (tumor burden occupying > 50% of liver)
* Major surgical procedure (as defined by the investigator) within 28 days prior to radioembolization. Note: Local surgery of isolated lesions for palliative intent is acceptable
* Participation in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 28 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or pharmacokinetics (PK) properties of an agent, a longer wash-out period will be required, as agreed by Regeneron and the investigator
* Prior exposure to anti-PD-1/PD-L1 inhibitor or anti-CTLA4 inhibitor, including cemiplimab in the past 12 months
* Any unresolved toxicity National Cancer Institute (NCI) CTCAE grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with cemiplimab may be included only after consultation with the study physician
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: Patients with vitiligo or alopecia; patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement; any chronic skin condition that does not require systemic therapy; patients without active disease in the last 5 years may be included but only after consultation with the study physician; patients with celiac disease that is controlled by diet alone
* History of allogeneic organ transplantation
* Expected radiation lung dose of > 30Gy
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study treatment and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of active primary immunodeficiency or acquired human immunodeficiency virus (HIV/AIDS)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study treatment. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment
* Active systemic infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice. Use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection
* History of leptomeningeal carcinomatosis
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Any concurrent chemotherapy, intraperitoneal (IP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
* Current or prior use of immunosuppressive medication within 14 days before the first dose of cemiplimab. The following are exceptions to this criterion: Intranasal, inhaled, topical steroid or local steroid injections (e.g., intra articular injection); systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent; steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 120 days (4 months) after the last dose of cemiplimab therapy or 120 days (4 months) days after the last TARE, whichever is longer
* Female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as per investigator discretion during the study. The rhythm method is not to be used as the sole method of contraception
* Male subjects, unwillingness to practice effective contraception (per Investigator discretion) while taking part in this study, because the effects of the SIR-Spheres treatment on sperm or upon the development of an unborn child are unknown
* Inability or unwillingness to understand or sign a written informed consent document
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* Presence of cardiovascular disease, as defined by:

  * New York Heart Association heart failure classifications of class II, III, or IV; or myocardial infarction, or acute coronary syndrome within 12 months of first dose of study medication; or
  * Transient ischemic attack or stroke within 1 year
* Any condition that requires ongoing/continuous corticosteroid therapy (> 10 mg prednisone/day or anti-inflammatory equivalent) within 1 week prior to the first dose of study medication. Participants who require a brief course of steroids (up to 2 days in the week before enrollment) or physiologic replacement are not excluded
* Ongoing or recent evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments
* Note: The following are not exclusionary: vitiligo, childhood asthma that has resolved, endocrinopathies (such as hypothyroidism or type 1 diabetes) that require only hormone replacement, or psoriasis that does not require systemic treatment
* Any infection requiring hospitalization or treatment with IV anti-infectives within 2 weeks of first dose of study medication
* Uncontrolled infection with HIV, hepatitis B or hepatitis C infection, diagnosis of immunodeficiency, and/or tuberculosis (active or latent)

  * Participants with known controlled HIV infection (undetectable viral load on HIV ribonucleic acid [RNA] polymerase chain reaction [PCR]) and CD4 count above 350 either spontaneously or on a stable antiviral regimen are eligible. For these participants monitoring will be performed per local standards
  * Participants with hepatitis B surface antigen (HBsAg) positive who have controlled infection (serum hepatitis B virus [HBV] deoxyribonucleic acid [DNA] PCR that is below the limit of detection and receiving anti-viral therapy for hepatitis B) are eligible. Participants with controlled infections must undergo periodic monitoring of HBV DNA. Participants must remain on anti-viral therapy for at least 6 months beyond the last dose of investigational study medication
  * Participants with HBsAg negative but total hepatitis B core antibody (HBcAb) positive are permitted with the following requirements: If serum HBV DNA PCR is above the limit of detection at screening, initiate HBV antiviral therapy before study entry. If serum HBV DNA PCR is below the limit of detection, periodic monitoring of HBsAg must be performed
  * Participants who are hepatitis C virus (HCV) antibody positive (Ab+) who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are eligible
* Receipt of a live vaccine within 4 weeks of start of study medication
* Receipt of COVID-19 vaccination within 1 week of planned start of study medication or for which the planned COVID-19 vaccinations would not be completed 1 week prior to start of study medication
* Known hypersensitivity to the active substances or to any of the excipients
* Women of childbearing potential (WOCBP) and men who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose. Highly effective contraceptive measures include:

  * Stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening;
  * Intrauterine device; intrauterine hormone-releasing system;
  * Bilateral tubal occlusion/ligation;
  * Vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has obtained medical assessment of surgical success for the procedure); and/or
  * Sexual abstinence
  * Pregnancy testing and contraception are required for WOCBP. Pregnancy testing and contraception are not required for women who are postmenopausal or permanently sterile
  * WOCBP are defined as women who are fertile following menarche until becoming postmenopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy
  * A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a postmenopausal state. The above definitions are according to the Clinical Trials Facilitation and Coordination Group (CTFG) guidance. Pregnancy testing and contraception are not required for women with documents hysterectomy or tubal ligation
  * Male participants: A male participant will be excluded from the study if that participant does not agree to use condoms or practice sexual abstinence, unless vasectomized, prior to the initial dose/start of study medication, during the study, and for at least 6 months after the last dose. Sperm donation is also prohibited during the same period. Vasectomy success must be confirmed by semen analysis
  * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drugs. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant
* Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
CD8+ T cell infiltration in tumor microenvironment (TME): baseline | At baseline
  Will be analyzed using multiplex immunofluorescence (IF) of formalin-fixed paraffin-embedded (FFPE) tissue. Will estimated the mean and standard deviation of the percent change.
CD8+ T cell infiltration in tumor microenvironment (TME): post TARE -1 (day 21) | At Post-transarterial radioembolization TARE -1 (day 21)
  Will be analyzed using multiplex immunofluorescence (IF) of formalin-fixed paraffin-embedded (FFPE) tissue. Will estimated the mean and standard deviation of the percent change.
CD8+ T cell infiltration in tumor microenvironment (TME): prior to TARE-2 (day 42) | At prior to TARE-2 (day 42)
  Will be analyzed using multiplex immunofluorescence (IF) of formalin-fixed paraffin-embedded (FFPE) tissue. Will estimated the mean and standard deviation of the percent change.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of study treatment
  Will be assessed and graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
T cell activation in TME: baseline | At baseline
  Will be analyzed using multiplex IF of FFPE.
T cell activation in TME: post-TARE-1 (day 21) | At Post-transarterial radioembolization TARE -1 (day 21)
  Will be analyzed using multiplex IF of FFPE.
T cell activation in TME: prior to TARE-2 (Day 42) | At prior to TARE-2 (Day 42)
  Will be analyzed using multiplex IF of FFPE.
Dendritic cell activation in TME: baseline | At baseline
  Will be analyzed using multiplex IF of FFPE.
Dendritic cell activation in TME: post-TARE-1 (day 21) | At Post-transarterial radioembolization TARE -1 (day 21)
  Will be analyzed using multiplex IF of FFPE.
Dendritic cell activation in TME: prior to TARE-2 (Day 42) | At prior to TARE-2 (Day 42)
  Will be analyzed using multiplex IF of FFPE.
PD-L1 expression in TME: baseline | At baseline
  Will be analyzed using multiplex IF of FFPE.
PD-L1 expression in TME: post-TARE-1 (day 21) | At Post-transarterial radioembolization TARE -1 (day 21)
  Will be analyzed using multiplex IF of FFPE.
PD-L1 expression in TME: prior to TARE-2 (Day 42) | At prior to TARE-2 (Day 42)
  Will be analyzed using multiplex IF of FFPE.
Immune activation | At baseline and post-TARE-1 (day 7-14)
  High parameter flow cytometry of peripheral blood samples used to assess proliferating (Ki-67+) CD8+ T cells, activated Tregs (CTLA-4+, TIGIT+), exhausted CD8+ T cells (PD-1high, CD39+, CD38+), CD8:Treg ratio, and myeloid derived suppressor cells (HLA-DR low monocytes).
Objective tumor response | Up to 2 years
  Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST (mRECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Kessler, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States